CLINICAL TRIAL: NCT07073716
Title: TAC, SOD and MDA Responses to Aerobic Exercise Versus Phoenix Seed in Obese Sedentary Females
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zainab Saeed Aly, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.T.REC/012/005432
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Aerobic Exercise Phoenix Seed, Antioxidant Potential
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise (Experimental): 20 subjects performed a specialized program of aerobic exercise with frequency of 3-5 times /week
  Interventions: Other: aerobic exercise
- phoenix seed (Experimental): 20 subjects performed specialized program of phoenix seed consumption
  Interventions: Dietary Supplement: phoenix seed
- Aerobic exercise and phoenix seed (Experimental): 20 subjects performed the same program of aerobic exercise with same frequency of 3-5 times /weeks combined with the same program of phoenix seed consumption
  Interventions: Combination Product: aerobic exercise+ phoenix seed

INTERVENTIONS:
Other: aerobic exercise — the exercise protocol was applied following these characteristics
  * frequency: 3-5 times /week along the whole study period
  * intensity: 70% of the maximal heart rate (220- age x 70/100)
  * duration: 50 min (warming up exercise movements (stretching and flexibility) in standing position, active phase of walking on a computerized treadmill, cooling down exercise movements (stretching and flexibility) performed in the seated position. being supervised by two trainers and the researcher. The researcher controlled the heartbeat 2 times through carotid pulse and At the end in order to restore the body to its initial state. all the patients could drink water during their training.
  Arms: Aerobic exercise
Dietary Supplement: phoenix seed — consuming 2 grams of phoenix seed powder dissolved in about 100 ml water 3 times/day
  Arms: phoenix seed
Combination Product: aerobic exercise+ phoenix seed — a specialized programme of aerobic exercise.the exercise protocol follow these characteristics
  * frequency: 3-5 times /week along the whole study period
  * intensity: 70% of the maximal heart rate (220- age x 70/100)
  * duration: 50 min (warming up exercise movements (stretching and flexibility) in standing position, active phase of walking on a computerized treadmill, cooling down exercise movements (stretching and flexibility) performed in the seated position. being supervised by two trainers and the researcher. The researcher controlled the heartbeat 2 times through carotid pulse and At the end in order to restore the body to its initial state. all the patients could drink water during their training.
  the specialized program of phoenix seed consumption (consuming 2 grams of phoenix seed powder dissolved in about 100 ml water 3 times/day)
  Arms: Aerobic exercise and phoenix seed

SUMMARY:
the aim of this study is To assess the antioxidant potential by measuring TAC, SOD and MDA responses to aerobic exercise versus phoenix seed in 60 obese sedentary females with symptoms of systemic inflammation. • All subjects will follow the given instructions strictly during the study duration, regarding the assessment and the treatment procedure, all participants will be evaluated under the same environmental conditions

DETAILED DESCRIPTION:
reactive oxygen species (ROS) are generated as metabolic by-products by biological systems during Processes like protein phosphorylation, activation of several transcriptional factors, apoptosis, immunity, and differentiation. When ROS production increases, they start showing harmful effects on important cellular structures like proteins, lipids, and nucleic acids. A large body of evidences shows that oxidative stress can be responsible, with different degrees of importance in the onset and/or progression of several diseases as cancer, diabetes, metabolic disorders, atherosclerosis, and cardiovascular diseases.

Date seed is a waste product that is high in polyphenolics (a mjor antioxidant compounds), phenolicacid (allergic, epicatechin, catechol,chlorogenic), carotenoids, total dietary fiber (such as pectin, β-glucan, and arabinoxylan), fat, protein, minerals, and various other nutrients and functional elements Phytosterols as β-sitosterol, campesterol, and Δ5-avenasterol are The major components of date seed oil sterols (contents varied between 4.70 and 8.45 mg/g) are important micronutrients and essential structural components of the cellular membrane.they serve crucial functions, such as modulating membrane permeability and fluidity, antioxidant activity , cholesterol-lowering effects and anti-inflammatory properties in addition to their putative contribution to reducing the risk of cardiovascular diseases and affording benefits to the immune system.

Physical activity improves antioxidant defences, lowers lipid peroxidation levels and involved in the protection from cardiovascular disorders, type II diabetes, metabolic syndrome and neurodegenerative diseases like Alzheimer's disease both in adult and in aged individuals. Thus emphasizing the importance of regular physical activity to decelerate the aging-associated impairment process.

Myokines,the bioactive peptides released by skeletal muscle following exercise as acrucial regulator of metabolic and protective pathways in peripheral tissues, particularly in combating oxidative stress and inflammation through activating intracellular signalling pathways within the liver that are involved in the liver's antioxidant defences.

this study aims to compare between aerobic exercise and phoenix seed in their antioxidant potential.

ELIGIBILITY:
Inclusion Criteria: sedentary obese female aged 35-55 years old with BMI of 30-39.9 and some symptoms of systemic inflammation (˃75 score at the inflammatory questionnaire) and had none of the exclusion criteria could be included in this study.

-

Exclusion Criteria: patients with orthopaedic or cardiac or any health condition that could interfere the ability to walk or exercise

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
TAC or total antioxidant capacity (blood test) | test applied before and after 2 months of the intervention protocol
  TAC: Determines the total antioxidant capacity of biological samples as a valuable approach to measuring health status under oxidative stress conditions,
SOD (superoxide dismutase) | Pre- intervention and after 8 weeks of treatment
  a blood test to determine the amount of SOD in blood and giving a good idea of the overall superoxide detoxifying capacity of a cell or tissue
MDA (malondialdehyde) | Pre- intervention and after 8 weeks of treatment
  blood test that measures Malondialdehyde (MDA) level as a marker of oxidative stress and a contributor to all major diseases by determining the impact of oxidation in normal and cancer cells.